CLINICAL TRIAL: NCT01785693
Title: Interest of a Bi-truncal Nerve Block (Femoral + Sciatic) Extended, Systematically Associated With General Anesthesia, in the Femoropopliteal Bypass: Study of Post-operative Analgesia and Peripheral Circulation Downstream.
Acronym: BLOC-FEMPOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: ARAMU Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-129; 2012-002123-15
Record Dates: First submitted 2013-01-17; First posted 2013-02-07 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Nerve block; Femoropopliteal bypass; Postoperative analgesia; Peripheral circulation; Levobupivacaine; Clonidine; Pain
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Pain | interventions — Levobupivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NaC1 (Other): The aim of this study is to assess, in patients scheduled for femoropopliteal bypass, the benefit of a double peripheral nerve block (femoral + sciatic) with levobupivacaine and clonidine in a single dose, performed before induction of general anaesthesia, on analgesia postoperatively assessed by morphine consumption.
  Interventions: Drug: levobupivacaine, clonidine
- Levobupivacaine + clonidine (Other): The aim of this study is to assess, in patients scheduled for femoropopliteal bypass, the benefit of a double peripheral nerve block (femoral + sciatic) with levobupivacaine and clonidine in a single dose, performed before induction of general anaesthesia, on analgesia postoperatively assessed by morphine consumption.
  Interventions: Drug: levobupivacaine, clonidine

INTERVENTIONS:
Drug: levobupivacaine, clonidine

SUMMARY:
The aim of this study is to assess, in patients scheduled for femoropopliteal bypass, the benefit of a double peripheral nerve block (femoral + sciatic) with levobupivacaine and clonidine in a single dose, performed before induction of general anaesthesia, on analgesia postoperatively assessed by morphine consumption.

Applied to the patient at the beginning of general anesthesia, this technique could allow one hand, to reduce the need for opiates, on the other hand - due to anesthetized limb vasodilation - to improve tissue perfusion downstream.

DETAILED DESCRIPTION:
Course of the study Visit 1 (J-15 J-1): Pre-inclusion During a follow-up visit usual pathology, the doctor will propose to the patient to participate in the protocol. Information Form will be given to the patient to be read at home to maintain a sufficient time for reflection.

Visit 2 (J-1): Pre-anesthetic, the eve of the intervention:

During the pre-anesthetic consultation routine, the doctor will check the informed consent and then note the following information on the case report form: age, height, weight, sex of the patient.

Visit 3 (J0): Surgery One hour before surgery the patient will receive premedication with Hydroxyzine (Atarax ®).

Then the anesthetic team install patient in monitoring room so that the test products are administered according to the double-blind randomization schedule prepared in advance. When the block is made, the patient is brought into the operating room for general anesthesia and surgery.

By the end of surgery, the following data will be collected in the case report form :

* Vital parameters (heart rate, blood pressure, PetCO2, SpO2) every 10 minutes and incidents.
* Time of injection tested products and time of induction of general anesthesia.
* Major Surgical times : incision, venous sampling when indicated, heparin bolus, clamping the superficial femoral artery, arterial unclamping, skin closure.
* Duration of operation (in minutes from the incision to skin closure).
* Intraoperative sufentanil consumption (micrograms).

Monitoring and medical care in Post Anaesthesia Carry Unit (PACU):

After surgery, the patient will be conducted in PACU. He will benefit from routine monitoring of vital parameters (heart rate, blood pressure, respiratory rate and SpO2).

Then patient extubation, according to usual criteria, will be performed: extubation of the patient is the H0, when all the time measurement start.

- H0: Extubation Morphine consumption will be measured continuously during the 72 first postoperative hours.

rSO2 be measured by NIRS during the first 12 first postoperative hours.

* H0 +30 min: rating of pain (simple numerical scale) + sedation score
* H0 +60 min: rating of pain + sedation score
* H0 +90 min: rating of pain
* H0 +120 min: rating of pain + sedation score
* H0+4h: rating of pain + sedation score
* H0+8h: rating of pain + sedation score
* H0+12h: rating of pain
* H0+16h: rating of pain + sedation score
* H0+20h: rating of pain
* H0+24h: rating of pain + sedation score + morphine consumption with PCA and number of requests over the last 24 hours.
* H0+32h: rating of pain
* H0+40h: rating of pain
* H0+48h: rating of pain + morphine consumption with PCA and number of requests over the last 24 hours.
* H0+56h: rating of pain
* H0+64h: rating of pain
* H0+72h: rating of pain + morphine consumption with PCA and number of requests over the last 24 hours.
* At the end of PACU: rating of pain + sedation score

Thereafter, recovery time of ambulation will be registered and duration of hospital stay, rate of reoperation within 30 post-operative days and 30-day survival.

Adverse events will be collected to have information about hemodynamic tolerance of the products.

The patient is then monitored in the usual care of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients to benefit a planned femoropopliteal bypass through PAOD stage II or III.
* Aged 18 to 80 years.
* Having given their consent.
* Affiliated with a social security scheme.

Exclusion Criteria:

* Patients with PAOD stage I or IV.
* Chronic respiratory failure.
* Severe coronary insufficiency.
* Renal or hepatic impairment.
* Patients with chronic pain or preoperative long-term opioid treatment.
* Patients with cognitive impairment (judged by the investigator) that may interfere with:

  * informed consent,
  * the collection of endpoints,
  * the use of patient-controlled analgesia.
* Severe abnormality of hemostasis (platelets <80.000 / ml) and / or of coagulation (PT <50%, factor V <50%).
* Patients with diabetes mellitus and / or diabetic neuropathy.
* Pregnant or nursing women, women of childbearing age.
* Refusal of the protocol.
* Minor or major protected patients.
* Contraindications to one of the following products:

levobupivacaine, clonidine, morphine, paracetamol, nefopam.

- Patients with a contra-indication to the administration of sufentanil: hypersensitivity to any component, hypersensitivity to morphine, hypersensitivity to opiates.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-01-30 (Actual); Primary Completion 2016-11-27 (Actual); Study Completion 2016-11-27 (Actual)

PRIMARY OUTCOMES:
total morphine consumption | between hour 0 and hour 0+24h

SECONDARY OUTCOMES:
total morphine consumption | between Hour 0 and Hour 0+72h
pain score at rest | 30, 60, 90 and 120 minutes after extubation
pain score | every 4 hours during the 24 first post-operative hours
pain score | every 8 hours during the next post-opeartive 48 hours
total sufentanil consumption | between induction and extubation
rate of reoperation | between day1 and day30
mortality rate | at day 30
sedation score | at hour0+30mn, at hour 0+1h, at hour 0+2h, at H0+4h, at hour 0+8h, at H0+16h, at hour 0+24h
Hemodynamic tolerance | between day 1 and day 30
nausea | between day 1 and day 30
vomiting | between day 1 and day 30
Bleeding score | between hour 0 and hour 0+24h

CONTACTS AND LOCATIONS:
Overall Officials: Philippe JOUVE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Charvin M, Longeras F, Jouve P, Cherprenet AL, Futier E, Pereira B, Duale C. Effects of adding a combined femoral and sciatic nerve block with levobupivacaine and clonidine to general anaesthesia in femoropopliteal bypass surgery: A randomised, double-blind, controlled trial. Eur J Anaesthesiol. 2020 Sep;37(9):787-795. doi: 10.1097/EJA.0000000000001263. PMID 32769505